CLINICAL TRIAL: NCT02021903
Title: Post-prandial Hypotension and Sleepiness in Parkinson's Disease and Other Synucleinopathies: the Model of an Oral Glucose Load
Brief Title: Post-prandial Hypotension and Sleepiness in Parkinson's Disease and Other Synucleinopathies
Acronym: HYPOSOMNPARK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 1120008
Record Dates: First submitted 2013-12-20; First posted 2013-12-27 (Estimated); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Parkinsonian Disorders
Keywords: arterial hypotension; postprandial sleepiness; orthostatic hypotension; synucleinopathies; hyperglycemia
MeSH Terms: conditions — Parkinsonian Disorders; Hypotension; Hypotension, Orthostatic; Synucleinopathies; Hyperglycemia | interventions — Meals

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HGPO + Placebo (Experimental): V1: HGPO 75 mg + meal and V2: Placebo 75 mg + meal
  Interventions: Other: V1: HGPO + meal and V2: placebo + meal
- Placebo + HGPO (Placebo Comparator): V1: Placebo 75 mg + meal and V2: HGPO 75 mg + meal
  Interventions: Other: V1: placebo 75mg + meal and V2: HGPO 75mg + meal

INTERVENTIONS:
Other: V1: HGPO + meal and V2: placebo + meal — * Ambulatory polysomnography for the night preceding each test
  * Usual antiparkinsonian treatments at their usual dose and timing
  * Randomisation to receive an oral solution of glucose load or a placebo (fructose). Standard meal 4 hours after the test
  * During two hours following the oral solution administration and the standardized meal, we will perform the followings for each patient :
    * continuous digital blood pressure monitoring by Nexfin®
    * blood pressure monitoring at brachial artery
    * continuous polysomnographic recording
    * synchronized continuous digital audiovisual recording
    * glucose and insulin blood level monitoring Additional blood samples will be taken in order to assay the intestine-pancreatic neuropeptides including incretins GLP- 1 and GIP
  Other Names: V1: HGPO 75mg + meal and V2: placebo 75mg + meal
  Arms: HGPO + Placebo
Other: V1: placebo 75mg + meal and V2: HGPO 75mg + meal — * Ambulatory polysomnography for the night preceding each test
  * Usual antiparkinsonian treatments at their usual dose and timing
  * Randomisation to receive an oral solution of glucose load or a placebo (fructose). Standard meal 4 hours after the test
  * During two hours following the oral solution administration and the standardized meal, we will perform the followings for each patient :
    * continuous digital blood pressure monitoring by Nexfin®
    * blood pressure monitoring at brachial artery
    * continuous polysomnographic recording
    * synchronized continuous digital audiovisual recording
    * glucose and insulin blood level monitoring Additional blood samples will be taken in order to assay the intestine-pancreatic neuropeptides including incretins GLP- 1 and GIP
  Arms: Placebo + HGPO

SUMMARY:
Excessive daytime sleepiness (EDS) is observed in 30 to 50 % of patients with Parkinson's disease (PD) patients, Dementia with Lewy Bodies (DLB) and Multiple System Atrophy (MSA). It is a major complain and represents a socially relevant problem as unintended episodes of sleep can also occur while driving for example. Arterial hypotension is frequently observed in patients with PD, DLB and MSA and considered as a marker of autonomic failure. Sleepiness is known to occur preferentially when patients are having arterial hypotension whatever the cause (i.e. postprandial period, administration of hypotensive medication such as dopamine agonists). We hypothesize that arterial hypotension is associated with abnormal sleepiness. We have observed this association in an on-going epidemiological survey Hyperglycaemia induced by oral glucose load - a standardized model simulating food intake during a meal - provokes arterial hypotension in the majority of Parkinson's disease patients with dysautonomia. It can be hypothesised that sleep attacks in these patients could be mediated by this fall in blood pressure.

DETAILED DESCRIPTION:
Excessive daytime sleepiness (EDS) is observed in 30 to 50 % of patients with Parkinson's disease (PD) patients, Dementia with Lewy Bodies (DLB) and Multiple System Atrophy (MSA). It is a major complain and represents a socially relevant problem as unintended episodes of sleep can also occur while driving for example. The exact pathophysiology of EDS in PD, DLB and MSA has not been fully elucidated so far, although pharmacological factors (dopaminergic medications) and pathological factors (neurodegeneration of sleep-wakefulness regulatory areas) have been identified. Arterial hypotension is frequently observed in patients with PD, DLB and MSA and considered as a marker of autonomic failure. Sleepiness is known to occur preferentially when patients are having arterial hypotension whatever the cause (i.e. postprandial period, administration of hypotensive medication such as dopamine agonists). We hypothesize that arterial hypotension is associated with abnormal sleepiness. We have observed this association in an on-going epidemiological survey (COPARK Cohort of 800 PD patients, manuscript in preparation). Hyperglycaemia induced by oral glucose load - a standardized model simulating food intake during a meal - provokes arterial hypotension in the majority of Parkinson's disease patients with dysautonomia. It can be hypothesised that sleep attacks in these patients could be mediated by this fall in blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Aged 35 to 85
* Parkinson's disease patients (UKPDSBB diagnostic criteria), patients with Dementia with Lewy Bodies (DLB consortium criteria, Mc Keith et al. 2005) or patients with Multiple System Atrophy (Gilman's criteria, 2008) complaining of a post-prandial sleepiness interfering with their daily living and with orthostatic hypotension
* Stable antiparkinsonian treatments (including those for dysautonomia) for the 2 months before the study and during the entire study
* Signed written informed consent for the present study
* Social security insurance coverage

Exclusion Criteria:

* atypical or secondary parkinsonism
* patients without excessive daytime sleepiness
* inability to give a consent due to severe cognitive dysfunction
* severe depression
* Deep brain stimulation treatment
* Moderate to severe obstructive sleep apnoea/hypopnoea syndrome or other co-morbidities that could account for abnormal daytime sleepiness
* Severe primary or secondary insomnia
* Treatment with sedative medications (unless moderate and stable treatment for more than 2 months before entering the study and maintained at stable dosage during all the study)
* Diabetes mellitus
* Systolic arterial pressure at rest in seated position lower than 100 mmHg in sitting position
* Pregnancy and suckling

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-05; Primary Completion 2019-12-20 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Rate of patients presenting a "sleep onset" | 2 hours
  Rate of patients presenting a "sleep onset", defined as the occurrence of at least 30 s of sleep at polysomnography or at patient's recall) with or without occurrence of hypotension (defined as a drop in systolic blood pressure level of at least 20 mmHg) during the 2 hours following oral glucose load or placebo fructose.

SECONDARY OUTCOMES:
rate of patients without arterial hypotension nor a sleep episode within 120 minutes after oral solution administration ; | 120 minutes
  rate of patients without arterial hypotension nor a sleep episode within 120 minutes after oral solution administration ;
rate of patients that show a sleep episode but without arterial hypotension within 120 minutes after oral solution administration ; | 120 minutes
  rate of patients that show a sleep episode but without arterial hypotension within 120 minutes after oral solution administration ;
rate of patients that show arterial hypotension within 120 minutes after oral solution administration but not a sleep episode; | 120 minutes
  rate of patients that show arterial hypotension within 120 minutes after oral solution administration but not a sleep episode;
Occurrence of arterial hypotension and a sleep episode within 120 minutes following a standardized meal | 120 minutes
  Occurrence of arterial hypotension (defined as a drop in systolic blood pressure level of at least 20 mmHg and a sleep episode (defined according to video-polygraphic parameters) within 120 minutes following a standardized meal (at lunch time)
Changes in intestine-pancreatic neuropeptides including incretins (GLP-1 - GIP) following an oral glucose load, placebo fructose load, or standardized meal - correlation with the post-prandial BP drop. | 120 minutes
  Changes in intestine-pancreatic neuropeptides including incretins (GLP-1 - GIP) following an oral glucose load, placebo fructose load, or standardized meal - correlation with the post-prandial BP drop.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Pavy-Le Traon, MD, Principal Investigator — University Hospital, Toulouse
Locations (2):
- France (2):
  - UHBordeaux, Bordeaux
  - UHToulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No